CLINICAL TRIAL: NCT00209625
Title: Phase I / II Study of Irinotecan (CPT-11) Combined With l-Leucovorin (l-LV) and 5-FU in Patients With Advanced Colorectal Cancer：Hokkaido Gastrointestinal Cancer Study Group:HGCSG0001
Brief Title: Phase I / II Study of Irinotecan (CPT-11) Combined With l-Leucovorin (l-LV) and 5-FU in Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hokkaido Gastrointestinal Cancer Study Group (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGCSG0001
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2000-04

CONDITIONS: Colorectal Cancer
Keywords: Irinotecan, leucovorin, fluorouracil, PhaseI/II, colorectal cancer,
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Leucovorin; Fluorouracil

INTERVENTIONS:
Drug: irinotecan
Drug: leucovorin
Drug: fluorouracil

SUMMARY:
We performed a phase I/II study of CPT-11/5FU/l-LV in advanced colorectal cancer, to determine the optimal dose of CPT-11 and to estimate the safety and efficacy of this regimen

DETAILED DESCRIPTION:
A multicenter Open-label, single-arm, phase I/II clinical trial is conducted on patients with histological stage IV colorectal cancer given irinotecan, leucovorin plus fluorouracil. The usefulness of this regimens as 1st line therapy for colorectal cancer was evaluated by the disease-free survival rate (DFR), median survival time (MST), incidence and severity of adverse event.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of colorectral adenocarcinoma.
2. Measurable or assessable lesions.
3. Age: 18 ~ 75 years.
4. Performance Status (ECOG): 0 ~ 2.
5. No prior chemotherapy. Adjuvant chemotherapy is not defined as previous therapy.
6. No history of radiotherapy to the abdomen.
7. Adequate function of major organs (bone marrow, heart, lungs, liver etc.). WBC 3,500/mm3 and 12,000/mm3. Hb 10.0 g/dl. Platelet count 100,000/mm3. GOT and GPT 2.5times the upper limit of normal (excluding liver metastasis). T-Bil 2.0mg/dl. Creatinine <1.5 mg/dl Normal ECG (not considering clinically unimportant arrhythmias and ischemic changes).
8. Predicted survival for >3 months.
9. Able to give written informed consent.

Exclusion Criteria:

1. Severe pleural effusion or ascites.
2. Metastasis to the central nervous system (CNS).
3. Active gastrointestinal bleeding.
4. Active infection.
5. Diarrhea (watery stools).
6. Uncontrolled ischemic heart disease.
7. Serious complications (such as intestinal paralysis, intestinal obstruction, interstitial pneumonia or pulmonary fibrosis, uncontrolled diabetes mellitus, heart failure, renal failure, or hepatic failure).
8. Active multiple cancer.
9. Severe mental disorder.
10. Pregnancy, possible pregnancy, or breast-feeding.
11. Flucytosine treatment
12. Gilbert's syndrome.
13. Judged to be ineligible for this protocol by the attending physician.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23
Dates: Start 2000-04; Study Completion 2004-11

PRIMARY OUTCOMES:
objective tumor response

SECONDARY OUTCOMES:
Response duration, time to progression, median survival time, and safety

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Asaka, MD, PhD, Study Chair — Hokkaido Gastrointestinal Cancer Study Group
Locations (1):
- Hokkaido University Hospital, Sapporo, Hokkaido, Japan